CLINICAL TRIAL: NCT05547841
Title: Normal Reference Value for Echocardiography in Chinese Han Pregnancies: a Prospective, Multicenter, Clinical Trial
Brief Title: Normal Reference Value for Echocardiography in Chinese Han Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: NO-REVAE-01
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; Echocardiography; Cardiac function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial group: A total of 680 singleton pregnant women in the first trimester (gestational age of 6-13 weeks + 6 days), who had normal results in various examinations and experienced regular obstetric examinations throughout the pregnancy, were selected from the obstetric outpatients in 34 centers, with 20 cases in each center.
  Interventions: Device: Echocardiography acquisition

INTERVENTIONS:
Device: Echocardiography acquisition — Echocardiography examination of all participants using PHILIPS. Time points for heart image acquisition in pregnant women: As per the Guidelines for Pre-pregnancy and Pregnancy Health Care (2018) formulated by the Obstetrics Group of the Gynecology Branch of the Chinese Medical Association, a total of six echocardiographic examinations will be performed in the first trimester (11-14 weeks of gestation), the second trimester(20-24 weeks of gestation), the third trimester (29-32 weeks of gestation), prenatal term (37-40 weeks of gestation), 6 weeks and 3-6 months after delivery. Time points for fetal heart image acquisition: Fetal heart images will be collected in the second trimester(20 to 24 weeks of gestation).

SUMMARY:
The First Hospital of China Medical University initiated a multi-center study on the reference range of echocardiography in Chinese Han Pregnancies to determine the reference range of echocardiography in the pregnant population and to promote the clinical application of echocardiography in the pregnant population, thereby offering the value of early evaluation and early diagnosis for cardiac structure and function in the pregnant population.

DETAILED DESCRIPTION:
During normal pregnancy, the cardiovascular system of pregnant women will undergo significant adaptive changes in response to the growth of the uterus, fetus and placenta. Cardiac output and plasma volume will increase by 40% to 50% compared with non-pregnancy. The heart rate continues to increase, while the blood pressure decreases in the first and second trimesters and increases in the third trimester. The heart structure of pregnant women also remodels during pregnancy and the inner diameter of the cardiac cavity and myocardial mass increase. The above changes usually return to pre-pregnancy levels within 3-6 months after delivery. Pregnancy can change hemodynamics and cardiac structure, thereby causing corresponding changes in maternal cardiac function.Therefore, it is very important to closely monitor the changes of pregnant women's cardiac structure and function during pregnancy to assess their adaptive changes.

In addition, the incidence of cardiovascular disease in pregnancy is 1-4% worldwide, and about 15% of maternal deaths are caused by complications related to cardiovascular diseases during pregnancy. In China, the proportion of maternal deaths caused by cardiovascular diseases during pregnancy is increasing yearly and cardiovascular diseases during pregnancy have become the primary cause of death for critically ill pregnant women. Previous studies have shown that common complications during pregnancy, such as gestational hypertension and diabetes, can also alter maternal heart function. Therefore, early detection of changes in left ventricular systolic function of pregnant women during pregnancy and after childbirth, timely treatment and early evaluation of treatment efficacy can greatly reduce their mortality.

Echocardiography is the preferred method for cardiac examination during pregnancy, because of its safe and convenient, and has no radiation risk to the mother and fetus. It can accurately and quickly measure and evaluate the size of the pregnant woman's heart cavity, hemodynamic changes and cardiac function, and reflect the adaptive changes. Continuous observation at different stages of pregnancy and postpartum can deeply reveal the changing of cardiac structure and function. However, due to the adaptive changes during pregnancy, the reference value of normal adult echocardiography cannot be directly applied to pregnant women in clinical practice. At present, there is still a lack of normal reference value of echocardiography for pregnancies in clinical practice.

In conclusion, in order to assess the cardiac changes of pregnancies more comprehensively and accurately, and find the pathological changes caused by cardiovascular diseases during pregnancy timely, it is urgent to establish the normal reference value of echocardiography in pregnancies. The purpose of this study is to establish the normal reference value range of echocardiography in Chinese Han pregnancies in different pregnancy periods and early postpartum period, and to explore the influencing factors of changes with gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Han nationality;
* 18-45 years old;
* Basal body mass index before pregnancy < 30 kg/m2;
* Normal blood pressure (139-90/89-60 mmHg);
* No history of cardiovascular and respiratory diseases;
* No abnormal findings in the physical examination of the cardiovascular and respiratory systems;
* Normal results in blood, urine, fasting blood glucose, blood lipids, liver and kidney function, thyroid function and electrocardiogram;
* Echocardiography shows normal cardiac function with no structural heart diseases;
* No use of medications that affect the cardiovascular system.

Exclusion Criteria:

* Anemia (hemoglobin < 90 g/L);
* Other serious diseases of the immune, respiratory, digestive, nervous, urinary, blood, endocrine and other systems;
* Tumors;
* The poor quality of ultrasound images cannot meet the requirements of parameter measurement and analysis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: A total of 680 singleton pregnant women in the first trimester, who had normal results in various examinations and experienced regular obstetric examinations throughout the pregnancy, were selected from the obstetric outpatients in 34 centers, with 20 cases in each center.
Sampling Method: Probability Sample
Enrollment: 680 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of echocardiographic parameters in Chinese Han pregnancies | From 11 weeks of gestation to 3-6 months postpartum
  To establish the normal reference range for echocardiography in Chinese Han pregnancies in different pregnancy periods.

SECONDARY OUTCOMES:
Measurement of left ventricular systolic and diastolic function using echocardiography | From 11 weeks of gestation to 3-6 months postpartum
  To establish the normal reference range of cardiac function for echocardiography in Chinese Han pregnancies in different pregnancy periods.

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, MD, Principal Investigator — First Hospital of China Medical University
Locations (34):
- China (34):
  - Chongqing Fifth People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Banan District People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Qianjiang District Central Hospital, Chongqing, Chongqing Municipality
  - Hainan Women and Children's Medical Center, Haikou, Hainan
  - Jiamusi Central Hospital, Jiamusi, Heilongjiang
  - Nanyang First People's Hospital, Nanyang, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Center Hospital of Wuhan, Wuhan, Hubei
  - Maternal and Child Health Care Hospital Hubei, Wuhan, Hubei
  - Jilin Provincial Women and Children Health Hospital, Changchun, Jilin
  - Jilin People's Hospital, Jilin, Jilin
  - Jilin Central General Hospital, Jilin, Jilin
  - Siping Women and Infants Hospital, Siping, Jilin
  - Yanji Maternal and Infant Hospital, Yanji, Jilin
  - Dalian Friendship Hospital, Dalian, Liaoning
  - Dalian Municipal Women and Children's Medical Center, Dalian, Liaoning
  - General Hospital of Fushun Mining Bureau, Fushun, Liaoning
  - Women And Children's Hospital of Jinzhou, Jinzhou, Liaoning
  - the First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shenyang Maternity And Child Health Hospital, Shenyang, Liaoning
  - Shenyang Women's and Children's Hospital, Shenyang, Liaoning
  - the First Hospital of China Medical Univeristy, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Tieling Women's And Children's Hospital, Tieling, Liaoning
  - Ningxia Maternal And Child Health Care Hospital, Yinchuan, Ningxia
  - Qinghai Provincial Maternal and Child Health Hospital, Xining, Qinghai
  - ShaanXi Province People's Hospital, Xi'an, Shaanxi
  - Heze Municipal Hospital, Heze, Shandong
  - Weifang Maternal and Child Health Hospital, Weifang, Shandong
  - ZiBo Central Hospital, Zibo, Shandong
  - Northwest Women's and Children's Hospital, Xi’an, Shanxi
  - Panzhihua Maternal and Child Hospital, Panzhihua, Sichuan
  - Yaan People's Hospital, Ya'an, Sichuan
  - Yunnan Maternal And Child Health Care Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided